CLINICAL TRIAL: NCT06958848
Title: Comparison of 16F Versus 24F Chest Drain After Minimally Invasive Pulmonary Lobectomy and/or Segmentectomy: a Monocentre Prospective Randomized Controlled Trial
Brief Title: 16F vs 24F Chest Drain After Minimally Invasive Lobectomy and/or Segmentectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-D0025; kt25Lardinois2
Record Dates: First submitted 2025-04-17; First posted 2025-05-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Pneumothorax; Pleural Effusion
Keywords: Lung Surgery; Chest Drainage; Minimally Invasive Thoracoscopic Lobectomy; Minimally Invasive Thoracoscopic Segmentectomy
MeSH Terms: conditions — Pneumothorax; Pleural Effusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 16F - early removal (Experimental): small-bore (16F) chest tubes, removal 2h until 6h after end of skin closure
  Interventions: Device: 16 F chest tube; Procedure: Early removal
- 16F - standard removal (Experimental): small-bore (16F) chest tubes, removal 1 day postoperative
  Interventions: Device: 16 F chest tube; Procedure: Standard removal
- 24F - early removal (Experimental): large-bore (24F) chest tubes, removal 2h until 6h after end of skin closure
  Interventions: Device: 24 F chest tube; Procedure: Early removal
- 24F - standard removal (Active Comparator): large-bore (24F) chest tubes, removal 1 day postoperative
  Interventions: Device: 24 F chest tube; Procedure: Standard removal

INTERVENTIONS:
Device: 16 F chest tube — Insertion of 16F chest tube
  Other Names: Small-bore chest tube
  Arms: 16F - early removal; 16F - standard removal
Device: 24 F chest tube — Insertion of 24F chest tube
  Arms: 24F - early removal; 24F - standard removal
Procedure: Early removal — Removal 2-6h after end of skin closure
  Arms: 16F - early removal; 24F - early removal
Procedure: Standard removal — Removal 1day postoperative
  Arms: 16F - standard removal; 24F - standard removal

SUMMARY:
The aim of the study is to evaluate postoperative pain in patients receiving a small-bore (16F) chest drain compared to those receiving the standard large-bore (24F) chest drain after minimally invasive pulmonary lobectomy and/or segmentectomy.

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related death worldwide, and surgical resection remains the treatment of choice for patients with resectable non-small cell lung cancer (NSCLC), particularly in early stages of the disease. Anatomical lung resections such as lobectomy and segmentectomy are commonly performed, increasingly through minimally invasive techniques like video-assisted thoracoscopic surgery (VATS) and robotic-assisted thoracoscopic surgery (RATS). Compared to traditional thoracotomy, VATS and RATS has been associated with better postoperative outcomes, including less pain, shorter hospital stays, faster recovery, and improved quality of life.

After lung resections, the standard postoperative management involves the insertion of a chest drain to remove air and fluid from the pleural space and monitor for complications such as air leaks or bleeding. Traditionally, most thoracic surgery centres use a single large-bore chest tube, typically 24F in size, which remains in place at least until the first postoperative day. However, this practice is not based on strong evidence, and there is currently no consensus on the optimal size of the chest drain. In fact, removal of the chest tube has been shown to significantly improve ventilatory function and reduce pain, particularly in the early postoperative period.

The Chest Drain 16F vs 24F Study investigates whether the use of a smaller-bore chest drain (16F) leads to less postoperative pain compared to the standard large-bore 24F drain in patients undergoing minimally invasive pulmonary lobectomy and/or segmentectomy. In addition to comparing the tube sizes, the trial explores the safety and feasibility of early chest drain removal, defined as removal within 2 to 6 hours after surgery, provided that specific clinical criteria are met (e.g., minimal air leak and no signs of complications). While retrospective data and small prospective studies suggest that early removal and the use of smaller tubes may be beneficial, high-quality prospective data are lacking. This study aims to provide evidence to potentially change clinical practice by reducing patient discomfort without compromising safety.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the patient (all sex and gender)
* Patients' age from ≥ 18 to ≤ 80 at time of study inclusion
* American Society of Anaesthesiologists (ASA) physical status classification I to III
* Patients with resectable non-small cell lung cancer (NSCLC) deemed operable by minimally invasive surgical technique (UICC Stages 0-II according to Tumor Nodes Metastasis (TNM) Classification 8th edition and selected patients with UICC Stage IIIA) or pulmonary metastasis or pulmonary lesion resected by lobectomy and/or segmentectomy
* Minimally invasive anatomical lung resections under general anaesthesia: lobectomy, lobectomy with wedge resection, lobectomy combined with segmentectomy, segmentectomy with wedge resection, bilobectomy

Exclusion Criteria:

* Previous thoracic surgery on the same side within 6 months
* Lung cancer complicated with pleural empyema
* Patients with chronic pain who receive opiates/gabapentin/pregabalin
* Patients who consume opiates/benzodiazepines
* Congestive heart failure NYHA Class III or IV
* Liver cirrhosis Child-Pugh Class B and C
* Renal insufficiency requiring dialysis and/or estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2
* Patients with coagulopathy or bleeding disorders: von Willebrand disease, Hemophilia; Thrombocytopenia (<50 G/l), requiring platelet transfusion
* Patients with neuralgia
* Chest pain (site of surgery) without taking painkillers, measured by VAS while coughing > 10 mm
* Rib fractures (in the last 3 months) on the side of surgical procedure
* Open anatomical lung resection, including pneumonectomy
* Insertion of 2 or more chest tubes
* Need for patient controlled intravenous anaesthesia or patient controlled epidural anaesthesia
* Patients intubated/sedated (not suitable due to difficulties to fill out the pain survey)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative chest pain | 2, 4 and 6 hours after last suture; twice daily from day 1 to day 3 postoperative or until tube removal; on discharge home, on follow up day 30 and 90
  Postoperative pain related to the placed chest drain (16F versus 24F), measured on a visual analogue scale (VAS) while coughing at different time points from skin closure until standard chest drain removal. The VAS is a horizontal line (100 mm) labelled from "no pain" on the left (0 mm) to "most extreme pain experienced" on the right (100 mm). Chest pain intensity is measured and recorded at rest and while coughing. For the current pain rating, the patient must be shown their last rating for comparison. The patient marks their information with a vertical line on the horizontal score line of the sheet paper. The evaluation is carried out by measuring the distance from the low anchor point to the marking; the recorded values are expressed in millimetres (0-100).
Postoperative acute pain relief while coughing | 2, 4 and 6 hours after last suture; twice daily from day 1 to day 3 postoperative or until tube removal; on discharge home, on follow up day 30 and 90
  Postoperative acute pain relief while coughing in the other 5 pairwise comparisons.
  Pain is measured on a visual analogue scale (VAS) while coughing. The VAS is a horizontal line (100 mm) labelled from "no pain" on the left (0 mm) to "most extreme pain experienced" on the right (100 mm).

SECONDARY OUTCOMES:
Postoperative acute pain relief at rest | 2, 4 and 6 hours after last suture; twice daily from day 1 to day 3 postoperative or until tube removal; on discharge home, on follow up day 30 and 90
  Postoperative acute pain relief at rest measured by an analgesia consumption adjusted pain intensity on a visual analogue scale at different time points in all subgroup comparisons. Pain is measured on a visual analogue scale (VAS) while coughing. The VAS is a horizontal line (100 mm) labelled from "no pain" on the left (0 mm) to "most extreme pain experienced" on the right (100 mm).
Analgesia consumption | 2, 4 and 6 hours after last suture; twice daily from day 1 to day 3 postoperative or until tube removal; on discharge home, on average up to 10 days postoperative; on 30- and 90 day follow up
  Intraoperative and postoperative analgesia consumption at different time points.
Duration of the thoracic drainage | From 2 until 6 hours post-surgery
  Duration of the thoracic drainage in hours from skin closure until chest tube removal if the air flow is ≤ 20 ml/min.
Fluid output | 2, 4 and 6 hours after last suture; twice daily from day 1 until discharge home, on average up to 10 days postoperative
  Duration of fluid output reported per 24h measured in ml/kg/24h with Medela Thopaz+™ until the chest tube is removed
Length of hospital stay | Patients are discharged from hospital on the 3rd to 7th day, or stay up to the 10th day in case of prolonged air leak or re-operation
  Length of hospital stay in nights from the end of the operation to the time when the patient is fit for discharge
Re-hospitalization | During hospitalization until 90-day follow-up
  Re-hospitalization due to pleural complications.
Postoperative morbidity | During hospitalization until 90-day follow-up
  Postoperative morbidity related to the medical device and/or procedure. Respiratory, thoracic, mediastinal and cardiac adverse events (AE). Adverse events are recorded and described according to CTCAE 5.0.
Pleural complications | During hospitalization until 90-day follow-up
  Pleural complications after early removal of chest tubes.The pleural complications will be graded according to Common Terminology Criteria for Adverse Events (CTCAE 5.0).
Mortality | During hospitalization, 30 and 90 days after hospital discharge
  In-hospital mortality; 30-day and 90-day mortality.
Chronic pain | 30 and 90 days after hospital discharge
  Chronic pain intensity and pain quality assessment while coughing and at rest on 30/90-day after hospital discharge.
Quality of life assessment | Preoperative, at hospital discharge and at 30/90-day follow-up
  Quality of life measured by Short Form 12 (SF-12) questionnaire. Score ranges from 0 to 100 while higher scores indicate better health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Didier Lardinois, MD, Study Chair — University Hospital, Basel, Switzerland; Makhmudbek Mallaev, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland